CLINICAL TRIAL: NCT04959383
Title: Exergame Balance Training for Pre Frontal Brain Activity and Executive Functioning in Patients With Mild Cognitive Impairment
Brief Title: Exergame Balance Training for Patients With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/1954 Aruba Saeed
Record Dates: First submitted 2021-06-26; First posted 2021-07-13 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Mild Cognitive Impairment
Keywords: Brain Activity; Executive Functions; Exergame balance training; Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low complexity Exergame balance training group (Experimental): Wobble board based exergame balance training, the game complexity will be low for this group.
  Interventions: Other: Low complexity Exergaming group
- Moderate complexity exergame balance training group (Experimental): Wobble board based exergame balance training, game complexity will be moderate for this group.
  Interventions: Other: Moderate complexity Exergaming group
- High complexity exergame balance training group (Experimental): Wobble board based exergame balance training, game complexity will be high for this group.
  Interventions: Other: High complexity Exergaming group
- Control group (Active Comparator): Wii fit based Exergame training on a stable surface
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Low complexity Exergaming group — This group will receive 30 minutes of Exergame Balance Training on Modified wobble board 3 times a week for 8 weeks. Wobble board will be able to rock in all direction with Weight Transfer. Wobble board based exergame balance training group game complexity will be kept low for this group.
  Other Names: Group A
  Arms: Low complexity Exergame balance training group
Other: Moderate complexity Exergaming group — This group will receive 30 minutes of Exergame Balance Training on Modified wobble board 3 times a week for 8 weeks. Wobble board will be able to rock in all direction with Weight Transfer. Wobble board based exergame balance training group game complexity will be kept moderate for this group.
  Other Names: Group B
  Arms: Moderate complexity exergame balance training group
Other: High complexity Exergaming group — This group will receive 30 minutes of Exergame Balance Training on Modified wobble board 3 times a week for 8 weeks. Wobble board will be able to rock in all direction with Weight Transfer. Wobble board based exergame balance training group game complexity will be kept high for this group.
  Other Names: Group C
  Arms: High complexity exergame balance training group
Other: Control Group — This group will receive 30 minutes of Exergame Balance Training on Modified wobble board 3 times a week for 8 weeks. This group will receive exergame balance training on Wii fit. Participants in this group will play Soccer Heading, Ski Slalom, Ski Jump, Table Tilt, Tightrope Walk, Balance Bubble, Penguin Slide and Snowboard Slalom game.
  Other Names: Group D
  Arms: Control group

SUMMARY:
This study will be a randomized control trial, which will be conducted on older adults with mild cognitive impairment. A specially designed Exergame balance training will be used for cognitive enhancement in patients with MCI. This training will determine the improvement in executive functioning, balance, speech and electrical activity of the brain.

DETAILED DESCRIPTION:
From last few years the line of research for cognitive enhancement has been shifted towards balance training as balance training is considered to directly stimulate the neuronal activity as compare to aerobic training. The previous finding also proposed that in aerobic training it is the intensity of training that improves the neuroplasticity and cognition but it is the neuro-cognitive demands and complexity of the task in balance training that affects the relationship between exercise and cognition in balance training. There is a need to determine the effect of the level of complexity of balance training on neural activity and executive functioning. Exergame augmented balance training is expected to have a better physical and cognitive outcome as compared to traditional balance training.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 55
* MoCA =20-24
* CDR ( dementia rating scale)≤ 1.0
* No unstable disease precluding planned exercise.
* Able to see and hear sufficiently to participate in planned physical and computer-based cognitive training.
* Patients score >45 on Berg Balance Scale.

Exclusion Criteria:

* Participation in any cognitive training activity
* Participation in > 150 min/wk of moderate or greater intensity planned exercise of any kind.
* Non-ambulatory or major mobility disorder.
* Other neurological conditions associated with cognitive impairment such as stroke, Parkinson disease, and head injury
* Any clinically significant psychiatric condition, current drug or alcohol abuse, or laboratory abnormality that would interfere with the ability to participate in the study.
* Individual with any musculoskeletal impairment.
* Unwillingness to participate.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Stroop test | 8th weeks
  Stroop test measure attention, processing speed, cognitive flexibility, and working memory. This test has good specificity (0.85-0.90). Coloured squares (red, green, blue) are presented in rows first (Stroop A), followed by those colour words typed in black ink (Stroop B), followed by incongruent colour words (Stroop C; in which participants will be asked to name the colour of the ink while ignoring the written word). A ratio will be computed to isolate the executive function component of the task. Assessment will be done at baseline, after the 4th and 8th week.
Trails Test | 8th weeks
  Trails test is used to assess selective attention, mental flexibility, visual-spatial skills and motor speed. It requires participants to connect numbered circles in ascending order. Color trails-2, requires individuals to connect numbered circles in consecutive order while also alternating the alphabets of the circle. Reliability and validity are adequate. Higher ratios represent a better executive function. Assessment will be done at baseline, after the 4th and 8th week.
Digit Span Forward and Backward | 8th weeks
  This test measures working memory's number storage capacity. It requires participants to first listen to a list of numbers and repeat them, with the string length increasing to the maximum of their ability. Digit Span Backward, requires repeating a string of numbers in reverse order. Continuing the pattern above to isolate the executive function component, the ratio of the typically smaller sum of correct interference trials on Digit Span Backward, divided by the typically greater sum of correct basic attention trials on Digit Span Forward. Assessment will be done at baseline, after the 4th and 8th week.
Montreal Cognitive Assessment | 8th weeks
  The MoCA was administered at baseline to characterize the sample as either normative aging or "screened as MCI" The MoCA consists of eight different subtests to assess overall cognitive impairment. Scores below 24 out of 30 were used to categorize MCI. This scale has a good reliability with Cronbach's alpha of 0.905. Its sensitivity is 88% and specificity is 98%. Assessment will be done at baseline, after the 4th and 8th week.
Alzheimer's disease Assessment Scale | 8th weeks
  Alzheimer's disease Assessment Scale will be used for Immediate and Delayed Recall Participants shows a list of 11 words on cards and they recall as many as they are able immediately and also after a delay interval. The number of errors/omissions comprises the score, so lower scores are better. It is a reliable tool with Cronbach's alpha of 0.83. Assessment will be done at baseline, after the 4th and 8th week.
Time Up and Go Test | 8th weeks
  The participants rise from sitting, walk 10 feet, turn around and return to the sitting position. The time it takes to complete the task is the score. Lower scores are better. It has a very good validity of 0.857. Assessment will be done at baseline, after the 4th and 8th week.
Mini Brief Balance Evaluation Systems | 8th weeks
  It is a reliable and valid tool. The mini Balance Evaluation Systems Test (BES Test) is a 14-item clinical balance assessment tool, developed to assess balance across six contexts of postural control: mechanical constraints, limits of stability, postural response to the induced loss of balance, sensory orientation, and gait. Assessment will be done at baseline, after the 4th and 8th week.
Smartphone Gait and Balance Application | 8th weeks
  The system consists of the following three components: i) a smartphone that has an embedded accelerometer, ii) a belt to house the phone on the lower back, iii) and a smartphone balance application. There are six different tasks that the subject have to perform with the system, like, normal walking up to 6 meters, walking with head movement, standing with eyes open and close and standing on a compromised surface with eyes open and close. This app. will calculate mediolateral and anterior-posterior sway during each task. Assessment will be done at baseline, after the 4th and 8th week.
Force Plate | 8th weeks
  Force Plate is a reliable and valid tool for balance assessment (ICC=0.8). In the force platform test, the mean velocity of the mediolateral (ML) and anterior-posterior (AP) movement of the COP will be calculated (mm/s) according to the displacement of the COP during each second. The mean moment of velocity (m m2/s) will be calculated as the mean of the areas covered by COP movement during each second of the Force Platform. Assessment will be done at baseline, after the 4th and 8th week.
Gait Speed Assessment | 8th weeks
  Self-selected gait speed (SSGS), fast gait speed (FGS), Cadence are considered to be decreased in patients with MCI. Gait speed will be assessed over 6 meters, and usual- and fast-pace walking mode. The test will be repeated twice with the mean of the two trials will be used for scoring purposes. Participants will be instructed to walk from a standing start at a pace that was normal and comfortable for them or to walk as fast as they could until they reached the end of the marked path. The participants will be asked to stop when their foot contacted the floor at the end of the walking course. Assessment will be done at baseline, after the 4th and 8th week.
Electroencephalography | 8th week
  An electroencephalography scalp electro-voltage activity (sampling frequency: 128Hz, bandpass hardware filter:1-32Hz) will be used. Delta, theta, beta1 and beta2 will be measured in eye open and closed state. Assessment will be done at baseline, after the 4th and 8th week.
Blood Biomarkers | 8th weeks
  The blood biomarkers will be assessed. A 5-mL blood sample will be obtained from the patient. The blood samples will be withdrawn for analysis of serum. The blood samples will be centrifuged. Samples will be and stored at - 80 °C for further serum marker assays. Assessment will be done at baseline, after the 4th and 8th week. Blood biomarkers BDNF, IGF-2, VEGF, TNFα, total-tau, amyloid beta-42, a-Synuclein, IL-10, IL1 and IL4 will be measured.

SECONDARY OUTCOMES:
Voice Recording | 8th weeks
  The Voice of all the patients will be recorded. Through voice recording pause length, verbal reaction time, and amount of silence will be assessed.
  Each participant performed four spoken tasks. The tasks consisted of a counting backward task, a sentence repeating task, an image description task, and a verbal fluency task. Each task will be recorded entirely to extract specific vocal features, including pause length, verbal reaction time, and amount of silence. Assessment will be done at baseline, after the 4th and 8th week.

OTHER OUTCOMES:
MRI of Brain | 8th weeks
  MRI Brain of patients will be carried out to evaluate the Gray matter volume in the hippocampus, prefrontal cortex, dorsolateral prefrontal cortex, the superior temporal sulcus and the anterior cingulate cortex. Assessment will be done at baseline, after the 4th and 8th week.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Amjad, PhD, Study Chair — Riphah international university.pakistan
Locations (1):
- Railway General Hospital, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fjell AM, Walhovd KB. Structural brain changes in aging: courses, causes and cognitive consequences. Rev Neurosci. 2010;21(3):187-221. doi: 10.1515/revneuro.2010.21.3.187. PMID 20879692
- [Background] Petersen RC, Doody R, Kurz A, Mohs RC, Morris JC, Rabins PV, Ritchie K, Rossor M, Thal L, Winblad B. Current concepts in mild cognitive impairment. Arch Neurol. 2001 Dec;58(12):1985-92. doi: 10.1001/archneur.58.12.1985. PMID 11735772
- [Background] Hanninen T, Hallikainen M, Tuomainen S, Vanhanen M, Soininen H. Prevalence of mild cognitive impairment: a population-based study in elderly subjects. Acta Neurol Scand. 2002 Sep;106(3):148-54. doi: 10.1034/j.1600-0404.2002.01225.x. PMID 12174174
- [Background] Angevaren M, Aufdemkampe G, Verhaar HJ, Aleman A, Vanhees L. Physical activity and enhanced fitness to improve cognitive function in older people without known cognitive impairment. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD005381. doi: 10.1002/14651858.CD005381.pub2. PMID 18425918
- [Background] Ludyga S, Gerber M, Brand S, Holsboer-Trachsler E, Puhse U. Acute effects of moderate aerobic exercise on specific aspects of executive function in different age and fitness groups: A meta-analysis. Psychophysiology. 2016 Nov;53(11):1611-1626. doi: 10.1111/psyp.12736. Epub 2016 Aug 24. PMID 27556572
- [Background] Saraulli D, Costanzi M, Mastrorilli V, Farioli-Vecchioli S. The Long Run: Neuroprotective Effects of Physical Exercise on Adult Neurogenesis from Youth to Old Age. Curr Neuropharmacol. 2017;15(4):519-533. doi: 10.2174/1570159X14666160412150223. PMID 27000776
- [Background] Christie BR, Eadie BD, Kannangara TS, Robillard JM, Shin J, Titterness AK. Exercising our brains: how physical activity impacts synaptic plasticity in the dentate gyrus. Neuromolecular Med. 2008;10(2):47-58. doi: 10.1007/s12017-008-8033-2. Epub 2008 Jun 6. PMID 18535925
- [Background] Fabre C, Chamari K, Mucci P, Masse-Biron J, Prefaut C. Improvement of cognitive function by mental and/or individualized aerobic training in healthy elderly subjects. Int J Sports Med. 2002 Aug;23(6):415-21. doi: 10.1055/s-2002-33735. PMID 12215960
- [Background] Barnes DE, Santos-Modesitt W, Poelke G, Kramer AF, Castro C, Middleton LE, Yaffe K. The Mental Activity and eXercise (MAX) trial: a randomized controlled trial to enhance cognitive function in older adults. JAMA Intern Med. 2013 May 13;173(9):797-804. doi: 10.1001/jamainternmed.2013.189. PMID 23545598
- [Background] Anderson-Hanley C, Arciero PJ, Brickman AM, Nimon JP, Okuma N, Westen SC, Merz ME, Pence BD, Woods JA, Kramer AF, Zimmerman EA. Exergaming and older adult cognition: a cluster randomized clinical trial. Am J Prev Med. 2012 Feb;42(2):109-19. doi: 10.1016/j.amepre.2011.10.016. PMID 22261206
- [Background] Hosseini SM, Kramer JH, Kesler SR. Neural correlates of cognitive intervention in persons at risk of developing Alzheimer's disease. Front Aging Neurosci. 2014 Aug 26;6:231. doi: 10.3389/fnagi.2014.00231. eCollection 2014. PMID 25206335
- [Background] Shubert TE, McCulloch K, Hartman M, Giuliani CA. The effect of an exercise-based balance intervention on physical and cognitive performance for older adults: a pilot study. J Geriatr Phys Ther. 2010 Oct-Dec;33(4):157-64. PMID 21717919
- [Background] Ries JD, Hutson J, Maralit LA, Brown MB. Group Balance Training Specifically Designed for Individuals With Alzheimer Disease: Impact on Berg Balance Scale, Timed Up and Go, Gait Speed, and Mini-Mental Status Examination. J Geriatr Phys Ther. 2015 Oct-Dec;38(4):183-93. doi: 10.1519/JPT.0000000000000030. PMID 25621384
- [Background] Rogge AK, Roder B, Zech A, Nagel V, Hollander K, Braumann KM, Hotting K. Balance training improves memory and spatial cognition in healthy adults. Sci Rep. 2017 Jul 18;7(1):5661. doi: 10.1038/s41598-017-06071-9. PMID 28720898
- [Background] Greblo Jurakic Z, Krizanic V, Sarabon N, Markovic G. Effects of feedback-based balance and core resistance training vs. Pilates training on cognitive functions in older women with mild cognitive impairment: a pilot randomized controlled trial. Aging Clin Exp Res. 2017 Dec;29(6):1295-1298. doi: 10.1007/s40520-017-0740-9. Epub 2017 Mar 1. PMID 28251569
- [Background] Eggenberger P, Wolf M, Schumann M, de Bruin ED. Exergame and Balance Training Modulate Prefrontal Brain Activity during Walking and Enhance Executive Function in Older Adults. Front Aging Neurosci. 2016 Apr 12;8:66. doi: 10.3389/fnagi.2016.00066. eCollection 2016. PMID 27148041
- [Background] Schattin A, Arner R, Gennaro F, de Bruin ED. Adaptations of Prefrontal Brain Activity, Executive Functions, and Gait in Healthy Elderly Following Exergame and Balance Training: A Randomized-Controlled Study. Front Aging Neurosci. 2016 Nov 23;8:278. doi: 10.3389/fnagi.2016.00278. eCollection 2016. PMID 27932975
- [Derived] Saeed A, Amjad I, Niazi IK, Alzahrani A, Shafiq M, Haavik H. Effects of Balance-Based Exergame Training With Variable Difficulty on Balance and Spatiotemporal Gait Outcomes in Adults With Mild Cognitive Impairment: Randomized Controlled Trial. JMIR Serious Games. 2025 Nov 18;13:e74092. doi: 10.2196/74092. PMID 41251404